CLINICAL TRIAL: NCT03649698
Title: Exercise and Nutrition for Healthy AgeiNg: Anabolic Interventions for Older People With (Pre)Sarcopenia to Improve Physical Functioning, Muscle Mass and Muscle Strength and to Understand the Underlying Mechanisms of Action.
Brief Title: Exercise and Nutrition for Healthy AgeiNg
Acronym: ENHANce
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); VISTA-Life (Unknown); Nestle Health Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S60763
Record Dates: First submitted 2018-08-07; First posted 2018-08-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Nutrition; Protein; Vitamin D; Exercise; Older people; Frailty
MeSH Terms: conditions — Sarcopenia; Motor Activity; Frailty | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * Participant: Yes blinded for protein and omega-3
  * Investigator: Yes blinded for protein and omega-3
  * Outcomes Assessor: Yes blinded for protein and omega-3
  * No blinding for exercise intervention.
  * Statistician is blinded for protein, omega-3 and exercise intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Home-based training program (Experimental): Home-based training program + protein placebo + omega-3 placebo
  Interventions: Behavioral: Home-based training program; Drug: Placebo protein powder; Drug: Placebo omega-3
- High-quality protein supplement (Experimental): High-quality protein supplement + omega-3 placebo
  Interventions: Dietary Supplement: High-quality protein supplement; Drug: Placebo omega-3
- 2 Anabolic interventions (Experimental): Home-based training program and high quality protein supplement
  Interventions: Behavioral: Home-based training program; Dietary Supplement: High-quality protein supplement; Drug: Placebo omega-3
- 3 Anabolic interventions (Experimental): Home-based training program, high-quality protein supplement and omega-3 fatty acids
  Interventions: Behavioral: Home-based training program; Dietary Supplement: High-quality protein supplement; Dietary Supplement: Omega-3 fatty acid
- Placebo protein powder and omega-3 (Placebo Comparator): Control group: protein placebo + omega-3 placebo
  Interventions: Drug: Placebo protein powder; Drug: Placebo omega-3

INTERVENTIONS:
Behavioral: Home-based training program — Exercise intervention: During the intervention period, the participant will perform the optimized and personally adapted Otago Exercise Program (OEP). The participant is encouraged to perform the resistance exercises three times a week with a rest day in between. The participant is advised to perform the exercises in close temporal proximity to one of the moments of the intake of the protein supplement. The participant will also follow a walking plan in which he or she needs to walk 30 minutes twice a week. These 30 minutes can be broken down to three 10-minute walks throughout the day. During the follow-up period, participants may continue the OEP, but no personal encouragement will be given during this period.
  Arms: 2 Anabolic interventions; 3 Anabolic interventions; Home-based training program
Dietary Supplement: High-quality protein supplement — The participant will receive an individually adapted protein supplement to achieve the recommend total (usual diet and supplements) daily intake of 1.5 g/protein/kg for frail elderly. This will be realized by adding an individualized amount (g) of protein powder during breakfast, lunch, dinner or snack between meals, or before breakfast or after dinner, based on the subjects' food intake assessed by a food diary. The participant will take the protein supplement from 5 days before the start of the intervention. The protein powder is commercially available and consists of 4.5g protein/5g powder. During the follow-up, no protein supplement is added.
  Arms: 2 Anabolic interventions; 3 Anabolic interventions; High-quality protein supplement
Dietary Supplement: Omega-3 fatty acid — Four weeks before the start of the intervention, the participant will start the intake of 1 omega-3 capsule providing in total 500 mg EPA and 450 mg DHA until the end of the intervention. He or she has to take the supplement once daily at a chosen time. During the follow-up, no omega-3 supplement will be given.
  Arms: 3 Anabolic interventions
Drug: Placebo protein powder — Isocaloric maltodextrin powder. Amount based on food diary.
  Arms: Home-based training program; Placebo protein powder and omega-3
Drug: Placebo omega-3 — Peanut oil soft gel capsules. 1g/ capsule. 1 capsule/day
  Arms: 2 Anabolic interventions; High-quality protein supplement; Home-based training program; Placebo protein powder and omega-3

SUMMARY:
The aim of this randomized placebo-controlled 5-arm clinical trial is to evaluate the effect of combined anabolic interventions compared to single or placebo interventions on physical performance in community-dwelling (pre)sarcopenic elderly (≥ 65 years) and to determine the underlying mechanisms of action. Important secondary outcome measures are muscle mass, muscle strength, compliance to the interventions (exercise program, protein and omega-3 supplementation) and functional, cognitive and nutritional status.

DETAILED DESCRIPTION:
The aim of this randomized 5-arm clinical trial is to evaluate the effect of combined anabolic interventions compared to single or placebo interventions on physical performance in community-dwelling (pre)sarcopenic elderly (≥ 65 years) living in Belgium. Physical performance will be evaluated using the Short Physical Performance Battery (SPPB). Muscle mass will be measured using a dual energy x-ray absorptiometry (DXA) and/or bioelectrical impedance analysis (BIA). Muscle strength will be measured by the Biodex (knee-extensor and knee-flexor) and a 1 hand-held dynamometer. The trial will also determine the underlying mechanisms of action using blood measures (such as markers of inflammation and sarcopenia) and muscle biomarkers. Important secondary outcome measures are compliance to the exercise program and to the protein and omega-3 supplementation, as well as functional, cognitive and nutritional status and the patients report on benefits and adverse events.

The study consists of four parts. Part I is the screening phase, which starts from the moment the participant has signed the informed consent until the start of the preparations of the study. During the screening, participants will be assessed for study eligibility by the study coordinator and contributors. If the participant is eligible, he or she will be randomly assigned into 1 of 5 intervention groups: Group 1: Exercise intervention; Group 2: Protein supplement; Group 3: Exercise intervention + protein supplement; Group 4: Exercise + Protein supplement + omega-3 supplement; Group 5: No intervention.

Part II is the preparation phase, in which the participants starts some of the interventions before the start of the study to familiarize patients with e.g. the intake of a protein supplement. All the participants will take an oral vitamin D supplement (800 IU cholecalciferol) from 4 weeks before the start of the intervention if their vitamin D level is above 20 nmol/L. Patients with a vitamin D level < 20 nmol/L will receive repletion therapy. A trial diary will be completed by all participants to record PA, falls and intake of protein/omega3/placebo and vitamin D products. Participants in the exercise intervention (group 1, 3 and 4) will be invited to an information session where the Otago Exercise Program (OEP) will be explained and practiced. With respect to the protein supplementation, participants will receive an individually adapted protein supplement to achieve the recommended total daily intake of 1.5 g protein/kg. This will be realized by adding an individualized amount (g) of protein powder during breakfast, lunch, dinner or snack between, before or after meals, based on the subjects' food intake assessed by a food diary. The protein powder is commercially available and consists of 4.5g protein/ 5g powder. The participants in group 2, 3 and 4 will start taking the protein supplement or matched placebo 5 days before the start of the intervention. Four weeks before the start of the intervention, the participants of group 4 will start with the intake of omega-3 (1 capsule providing in total 500 mg eicosapentanoic acid (EPA) and 450 mg docosahexaenoic acid (DHA)) or matched placebo. Placebo will be provided for the participants who are not given a protein and/or omega-3 supplement. Participants are blinded to the nutritional interventions.

The third part of the study, the intervention period, takes 12 weeks. During this period, there are 8 contact moments (at baseline, week 1, week 2, week 4, week 6, week 8, week 10 and week 12). All the participants continue with the vitamin D supplementation. Participants in the exercise intervention (group 1, 3 and 4) will perform the optimized and personally adapted OEP and will also follow a walking plan. The strength exercises of the OEP are personalised based on the individual's 1 repetition maximum. Balance exercises of the OEP are personalised based on improvements on MiniBESTest scores during the intervention period. The nutritional intervention groups (protein supplementation: group 2, 3 and 4 and omega-3 supplementation: group 4) continue with the protein and/or omega-3 supplements until the last visit of the intervention period.

Part IV is the follow-up period, after the intervention. This phase takes 12 weeks and exists of 2 telephone contacts and 2 contact moments. All the participants continue the vitamin D supplementation until the last visit of the follow-up. The exercise intervention group (group 1, 3 and 4) may continue the OEP, but no personal encouragement will be given during this period. No protein and/ or omega-3 supplements will be given during the follow-up.

Several outcomes will be measured during the contact moments of the intervention period and follow-up period (part III and part IV). This will be done by questionnaires about nutritional status, fall history and use of health care (from baseline until end of follow-up), and evaluation of functional and cognitive status. Blood, urine and muscle samples will be taken. The physical activity will be measured by wearing a movement tracker. All participants will wear a movement tracker 5 days before the intervention period and during the first two weeks of the intervention period and last two weeks of the intervention period, and during the last 2 weeks of the follow-up period. Participants who receive an exercise intervention (group 1, 3 and 4) will be encouraged to wear the movement tracker during the complete intervention period. The participants will complete a four-day food diary throughout the trial at week 1, week 6, week 12 and week 24. The participants will be asked for compliance during the preparation period and intervention period and their fall history which can be monitored by using diaries during the intervention period and the follow-up period.

Addendum 27-07-2021: starting from 01-2021 a substudy was initiated in which participants of ENHANce, who agreed for participation in this substudy, collect stool samples at baseline, week 4, week 8 and week 12 of the intervention. This will allow to observe possible changes in gut microbiota composition and intestinal inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female persons with (pre)sarcopenia according to the European Working Group on Sarcopenia in Older People (EWGSOP): reduced muscle mass without (presarcopenia) or with (sarcopenia) reduced walking speed (≤ 0.8m/s) or muscle strength OR probable, confirmed or severe sarcopenia according to EWGSOP 2.
2. 65 years or older;
3. Community-dwelling elderly or assisted living;
4. In case of one or more positive answer(s) on the health screen for exercise, subjects need approval of their general practitioner to participate in this randomized controlled trial (RCT).

   * Uncontrolled or unstable health problems
   * Uncontrolled pain or feeling unwell the day of the exercise
   * Recently diagnosed cardiovascular events
   * systolic blood pressure (SBP) ≥ 180 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mmHg
   * Resting tachycardia > 100 bpm
   * Uncontrolled atrial or ventricular arrhythmias
   * Unstable or acute heart failure
   * Lasting, increased pain following a previous session
   * Suspected acute injury
   * Recent injurious fall without medical assessment
   * Severe breathlessness or dizziness
   * Uncontrolled pulmonary problems
   * Rheumatoid arthritis flare up or acute systemic illness/infection
   * Unexplained lethargy

Exclusion Criteria:

1. Impairments/diseases that impose problems to participation in the study;
2. Allergy to milk or soy or peanut;
3. Mini-Mental State Examination (MMSE) < 21;
4. Terminal illness (prognosis < 6 months);
5. Persons who followed a physical training program in the last 6 months (twice or more/week);
6. Persons with a daily intake of > 1.5 g protein/kg body weight (BW)/day;
7. Diagnosis of severe kidney disease (GFR < 30 ml/min) or diabetes mellitus;
8. Unable to communicate in Dutch, English or French.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-02-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change in physical functioning | Measured at baseline, week 12 and week 24.
  Change in SPPB score
Percentage of participants with change in physical functioning | Measured at baseline, week 12 and week 24.
  the percentage of participants with more than 1 or 1 point increase in SPPB score.

SECONDARY OUTCOMES:
Change in muscle mass (after intervention-baseline) | Measured at screening, week 12 and week 24 with DXA or when screening is 6 weeks prior to baseline, DXA will also be performed at baseline. At screening, baseline, week 12 and week 24 with BIA.
  Appendicular lean mass will be measured with a whole-body DXA scan and by BIA.
Change in muscle strength (after intervention-baseline) | Hand grip measured at screening, baseline, week 12 and week 24. Biodex measured at baseline, week 12 and week 24.
  Muscle strength of the knee-extensor, knee-flexor and hip abductors will be measured by Biodex and hand grip strength with dynamometer.
Compliance to the exercise intervention, subjective | baseline until week 12
  Compliance to the Otago program will be assessed by measure of:
  - The number of Otago sessions the participant performed divided by the number of Otago sessions the participants needed to perform. Likewise, this will be calculated for the walking program and for the integral exercise intervention.
Compliance to the exercise intervention, objective | baseline until week 12
  Compliance to the Otago program will be assessed by measure of:
  - Monitor and diary: Length of exercise session (time). Pattern recognition of exercise groups by algorithm development
Compliance to the exercise intervention, subjective, detailed | baseline until week 12
  Compliance to the Otago program will be assessed by measure of:
  - Diary: the reported intensity of the strength exercises
Compliance to the protein supplementation, objective | Urine samples at baseline, week 1, 2, 4, 6, 8, 10, 12, 24.
  Compliance to protein supplementation:
  - The number of nutritional intakes the participant did divided by the number of intakes of nutritional supplement the participant was prescribed.
Compliance to the protein supplementation, subjective | Urine samples at baseline, week 1, 2, 4, 6, 8, 10, 12, 24.
  Compliance to protein supplementation:
  - Count and weight returned powder boxes
Compliance to the protein supplementation objective | Urine samples at baseline, week 1, 2, 4, 6, 8, 10, 12, 24.
  Compliance to protein supplementation:
  - N content in 8 24h urine samples by the Dumas method (28) to estimate rise in protein intake and Creatinine index to estimate the completion of the urine samples (29, 30)
Compliance to the omega-3 supplementation, subjective | baseline, week 12 and week 24.
  Compliance to omega-3 supplement
  - Count returned capsules and placebo tablets
Compliance to the omega-3 supplementation, objective | baseline, week 12 and week 24.
  Compliance to omega-3 supplement
  - Compliance to the omega- 3 supplement is assessed by counting the number of capsules during each study visit and by analysis of red blood cell (RBC) membrane fatty acid profile
Functional status: frailty | baseline, week 12 and 24
  - Change in physical frailty stage defined by Fried et al (frail (3-5/5), prefrail (1-2/5), robust (0/5))
Functional status: activities of daily living | baseline, week 12 and 24
  Change in activity of daily living (ADL) :Barthel-index
Functional status: balance | baseline, week 12 and 24
  Change in balance (Mini-BESTest)
Functional status: change in physical activity | baseline, week 12 and 24
  Change in PA by the MoveMonitor+ (MM+) (method under development in our research group)
Functional status: health-related quality of life | baseline, week 12 and 24
  - Change in health-related quality of life, according to Short Form Health Survey (SF-36) questionnaire
Functional status: falls | baseline, week 12 and 24
  - Number of falls and the circumstances, identified using weekly fall calendars + Falls Efficacy Scale International (FES-I)
Cognitive status: immediate and delayed memory, attention, language and visuospatial skills | baseline, week 12 and 24
  - The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): immediate and delayed memory, attention, language and visuospatial skills;
Cognitive status: inhibition | baseline, week 12 and 24
  Stroop test (inhibition)
Cognitive status | baseline, week 12 and 24
  - Maze test
Nutritional status: malnutrition | at baseline (preparation for food diary), week 6, week 12 and week 24
  - Changes in numbers of participants with malnutrition, according to Mini Nutritional Assessment (MNA).
Nutritional status: nutrient intake | at baseline (preparation for food diary), week 6, week 12 and week 24
  - Changes in nutrient intake, according to the four day food diary.
Patient reported benefits and adverse effects | week 1, 4, 8, 12, 16, 20, 22, 24.
  Benefits and adverse effects are asked. Participants will describe their thoughts about the study, what they like and don't like.
Change in C reactive protein (CRP) | baseline, week 1, 4, 12 and 24
  change in hs-CRP
Change in hemoglobin | baseline, week 12 and week 24
  Change in hemoglobin
Change in creatinine | baseline, week 12 and week 24
  Change in creatinine
Change in urea | baseline, week 12 and week 24
  Change in urea
Change in serum albumin | baseline, week 12 and week 24
  Change in serum albumin
Change in glucose | baseline, week 12 and week 24
  Change in glucose
Change in cholesterol (HDL, LDL, total, Triglycerides) | baseline, week 12 and week 24
  Change in cholesterol (HDL, LDL, total, Triglycerides)
Change in insulin | baseline, week 12 and week 24
  Change in insulin
Change in insulin like growth factor 1 (IGF-1) | baseline, week 12 and week 24
  Change in IGF-1
Change in 25-hydroxy-vitamin D | baseline, week 12 and week 24
  Change in 25-hydroxy-vitamin D
Change in creatinine kinase | baseline, week 12 and week 24
  Change in creatinine kinase
Change in indoxyl sulfate | baseline, week 12 and week 24
  Change in indoxyl sulfate
Change in interleukin 6 (IL-6) | baseline, week 12 and week 24
  Change in IL-6
Change in IL-1b | baseline, week 12 and week 24
  Change in IL-1b
Change in tumor necrosis factor alpha (TNF-alpha) | baseline, week 12 and week 24
  Change in TNF-alpha
Change in myostatin | baseline, week 12 and week 24
  Change in myostatin
Change in activin A | baseline, week 12 and week 24
  Change in activin A
Change in markers of muscle wasting | baseline, week 12
  Change in markers of muscle wasting (MURF1, Atrogin1, FOXO3)
Change in markers of muscle regeneration | baseline, week 12
  Change in markers of muscle regeneration (PAX7, Myogenic factor 5 (MYF5), myoblast determination protein (MyoD), Ki67, mammalian target of rapamycin (mTOR), AMPK)
Change in muscle histology | baseline, week 12
  Change in muscle histology
Change in composition of gut microbiota | baseline, week 4, week 8, week 12
  Change in composition of gut microbiota
Change in markers of intestinal inflammation | baseline, week 4, week 8, week 12
  Change in markers of intestinal inflammation (fecal calprotectin, lactoferrin, S100A12)

CONTACTS AND LOCATIONS:
Overall Officials: Evelien Gielen, Prof MD PhD, Principal Investigator — Gerontology and Geriatrics, Department of Public Health and primary care KU Leuven
Locations (1):
- Gerontology and Geriatrics, Department of Public Health and Primary Care, KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Amini N, Dupont J, Lapauw L, Vercauteren L, Peeters L, Dedeyne L, Verschueren S, Tournoy J, Gielen E. A multicomponent intervention consisting of exercise, proteins and omega-3 supplementation to improve sarcopenia in community-dwelling older adults: Lessons learned from a 5-armed randomized controlled feasibility trial. J Frailty Aging. 2026 Feb 2;15(1):100129. doi: 10.1016/j.tjfa.2025.100129. Online ahead of print. PMID 41632571
- [Derived] Amini N, Devriendt A, Lapauw L, Dupont J, Vercauteren L, Verbeke K, Verschueren S, Tournoy J, Gielen E. Estimating protein intake in sarcopenic older adults: combining food diaries and weighed powders versus 24-hour urine collections. J Nutr Health Aging. 2025 Mar;29(3):100474. doi: 10.1016/j.jnha.2024.100474. Epub 2025 Jan 8. PMID 39787986
- [Derived] Lapauw L, Dupont J, Amini N, Vercauteren L, Verschueren S, Tournoy J, Raes J, Gielen E. Trial in Elderly with Musculoskeletal Problems due to Underlying Sarcopenia-Faeces to Unravel the Gut and Inflammation Translationally (TEMPUS-FUGIT): protocol of a cross-sequential study to explore the gut-muscle axis in the development and treatment of sarcopenia in community-dwelling older adults. BMC Geriatr. 2023 Sep 26;23(1):599. doi: 10.1186/s12877-023-04291-5. PMID 37752426
- [Derived] Dedeyne L, Dupont J, Koppo K, Verschueren S, Tournoy J, Gielen E. Exercise and Nutrition for Healthy AgeiNg (ENHANce) project - effects and mechanisms of action of combined anabolic interventions to improve physical functioning in sarcopenic older adults: study protocol of a triple blinded, randomized controlled trial. BMC Geriatr. 2020 Dec 10;20(1):532. doi: 10.1186/s12877-020-01900-5. PMID 33302879